CLINICAL TRIAL: NCT02669433
Title: A Phase 2b, Double-Blind, Randomized, Placebo-Controlled Study of RVT-101 in Subjects With Dementia With Lewy Bodies (DLB)
Brief Title: Study Evaluating Intepirdine (RVT-101) in Subjects With Dementia With Lewy Bodies: The HEADWAY-DLB Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Axovant Sciences Ltd. (Industry)
Responsible Party: Sponsor
Organization: Sio Gene Therapies (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RVT-101-2001
Record Dates: First submitted 2016-01-25; First posted 2016-02-01 (Estimated); Results first posted 2019-04-26 (Actual); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Dementia With Lewy Bodies
Keywords: Dementia with Lewy bodies; Lewy bodies; intepirdine; RVT-101; dementia
MeSH Terms: conditions — Lewy Body Disease; Dementia | interventions — 3-benzenesulfonyl-8-piperazin-1-ylquinoline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- RVT-101 35 mg (Experimental): RVT-101 35 mg once daily
  Interventions: Drug: RVT-101 35 mg
- RVT-101 70 mg (Experimental): RVT-101 70 mg once daily
  Interventions: Drug: RVT-101 70 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RVT-101 35 mg — once daily, oral, 35-mg tablets
  Arms: RVT-101 35 mg
Drug: RVT-101 70 mg — once daily, oral, 35-mg tablets
  Arms: RVT-101 70 mg
Drug: Placebo — once daily, oral, matching tablets
  Arms: Placebo

SUMMARY:
This study seeks to evaluate the efficacy and safety of intepirdine (RVT-101) in patients with dementia with Lewy bodies.

DETAILED DESCRIPTION:
The efficacy and safety of RVT-101 at doses of 70 mg and 35 mg daily will be evaluated over a 24-week double-blind treatment period in patients with dementia with Lewy bodies.

The randomization ratio will be 1:1:1 (70 mg RVT-101: 35 mg RVT-101: placebo).

Subjects completing this study will be eligible to enroll in an extension study of RVT-101 (Study RVT-101-2002).

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject with probable DLB
* Mini Mental State Examination (MMSE) score of 14-26 inclusive at Screening and Baseline
* Patient has the ability to comply with procedures for cognitive and other testing in the opinion of the investigator
* Patient has a reliable caregiver who is willing to report on the subject's status throughout the study
* Patients currently receiving therapy for DLB are eligible for enrollment

Exclusion Criteria:

* Atypical clinical features or clinical course that would lead the investigator to conclude primary symptoms are more likely explained by an alternate dementia diagnosis.
* Any clinically relevant concomitant disease that, in the opinion of the investigator, makes the patient unsuitable for inclusion in the study.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ilise Lombardo, MD, Study Director — Axovant Sciences Inc., Senior Vice President, Clinical Research
Locations (65):
- United States (31):
  - US138, Phoenix, Arizona
  - US108, Phoenix, Arizona
  - US139, Sun City, Arizona
  - US125, Tucson, Arizona
  - US119, Irvine, California
  - US134, Oxnard, California
  - US133, Rancho Mirage, California
  - US140, Sacramento, California
  - US141, Englewood, Colorado
  - US123, Washington D.C., District of Columbia
  - US104, Boca Raton, Florida
  - US116, Boca Raton, Florida
  - US111, Jacksonville, Florida
  - US122, Orlando, Florida
  - US137, Palm Beach Gardens, Florida
  - US126, Tampa, Florida
  - US136, Atlanta, Georgia
  - US112, Chicago, Illinois
  - US118, Indianapolis, Indiana
  - US105, Lexington, Kentucky
  - US135, Newton, Massachusetts
  - US130, Quincy, Massachusetts
  - US102, Rochester, Minnesota
  - US109, New York, New York
  - US100, Chapel Hill, North Carolina
  - US110, Cleveland, Ohio
  - US106, Columbus, Ohio
  - US131, Portland, Oregon
  - US120, Willow Grove, Pennsylvania
  - US124, Dallas, Texas
  - US101, Charlottesville, Virginia
- Canada (2):
  - CA200, Toronto, Ontario
  - CA201, Sherbrooke, Quebec
- France (10):
  - FR952, Toulouse, Haute-Garonne
  - FR957, Lille, Nord
  - FR951, Villeurbanne, Rhône
  - FR954, Bron
  - FR959, Paris
  - FR956, Paris
  - FR960, Paris
  - FR953, Saint-Herblain
  - FR950, Strasbourg
  - FR955, Vandœuvre-lès-Nancy
- Italy (6):
  - IT304, Tricase, Lecce
  - IT300, Genoa, Liguria
  - IT302, Brescia, Lombardy
  - IT306, Brescia
  - IT301, Milan
  - IT305, Venice
- Netherlands (3):
  - NE402, Amsterdam, North Holland
  - NE401, 's-Hertogenbosch
  - NE400, Rotterdam
- Spain (3):
  - SP600, Barcelona
  - SP605, Barcelona
  - SP602, Burgos
- United Kingdom (10):
  - UK801, Cambridge, Cambridgeshire
  - UK808, Epping, Essex
  - UK804, Southampton, Hampshire
  - UK807, Bristol
  - UK806, Dundee
  - UK805, Isleworth
  - UK800, London
  - UK809, London
  - UK802, Manchester
  - UK803, Newcastle upon Tyne

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 484 participants signed consent and were screened for participation. Of these, 306 entered a 2-week single-blind placebo run-in period with treatment with placebo qd. There was an overlap between the participants from the run-in period and the participants that were randomized during the treatment period.
Groups:
- Placebo: Subjects dosed with two Placebo tablets
  Placebo: once daily, oral, matching tablets
- RVT-101 35 mg: Subjects dosed with one Placebo tablet + 1 35 mg tablet of RVT-101
  RVT-101 35 mg: once daily, oral, 35-mg tablets
- RVT-101 70 mg: Subjects dosed with two RVT-101 35 mg tablets
  RVT-101 70 mg: once daily, oral, 35-mg tablets
Period: Overall Study
Arm/Group | Placebo | RVT-101 35 mg | RVT-101 70 mg
Started | 91 | 89 | 89
Safety Population (The Safety population included subjects who took at least 1 dose of double-blind study drug) | 91 | 89 | 88
Intent to Treat (ITT) Population (Subjects took at least 1 dose of double-blind study drug and had at least 1 post-baseline assessment) | 89 | 89 | 87
Per-Protocol Population (Subjects in the ITT population who had no major protocol violations) | 78 | 79 | 82
Completers Population (Subjects in the ITT population who completed the study) | 73 | 72 | 69
UPDRS Primary Population | 87 | 87 | 84
Completed (Subjects who completed every visit per protocol) | 76 | 75 | 74
Not Completed | 15 | 14 | 15
Not completed — Protocol Violation | 0 | 4 | 1
Not completed — Disease Progression | 1 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0
Not completed — Adverse Event | 6 | 7 | 10
Not completed — Sponsor Termination | 1 | 0 | 1
Not completed — Withdrawal by Subject | 5 | 1 | 0
Not completed — Withdrawal by Caregiver | 1 | 0 | 2
Not completed — Death | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | RVT-101 35 mg | RVT-101 70 mg | Total
Number analyzed (Participants) | 91 | 89 | 88 | 268
Age, Continuous [Mean (Full Range); unit: years] | 73.6 [59 to 86] | 73.0 [55 to 85] | 73.0 [55 to 86] | 73.0 [55 to 86]
Age, Customized [Count of Participants; unit: Participants]
  < 74 years | 45 | 45 | 45 | 135
  >/= 74 years | 46 | 44 | 43 | 133
  < 65 years | 7 | 9 | 12 | 28
  >/=65 years | 84 | 80 | 76 | 240
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 22 | 15 | 57
  Male | 71 | 67 | 73 | 211
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 0 | 10
  Not Hispanic or Latino | 86 | 83 | 86 | 255
  Unknown or Not Reported | 1 | 0 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 3 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 4 | 0 | 4
  White | 90 | 81 | 85 | 256
  More than one race | 0 | 1 | 0 | 1
  Unknown or Not Reported | 1 | 0 | 2 | 3
BMI [Mean (Full Range); unit: kg/m^2] — Population: Data was missing for two subjects
  kg/m^2
    number analyzed (Participants) | 90 | 89 | 87 | 266
    (all) | 26.59 [15.8 to 39.2] | 26.51 [16.8 to 42.1] | 26.81 [18.6 to 41.6] | 26.64 [15.8 to 42.1]

OUTCOME MEASURES:

1. Primary Outcome: Unified Parkinson's Disease Rating Scale-Part III (UPDRS-III) Change From Baseline at Week 24
Description: The primary endpoint was to assess the effects of intepirdine versus placebo on the UPDRS Part III after 24 weeks of treatment. UPDRS Part III scores range from 0 to 108, with higher scores indicating worse outcome.
Time Frame: Change from Baseline at 24 weeks
Population: UPDRS Primary Population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | RVT-101 35 mg | RVT-101 70 mg
Number analyzed (Participants) | 72 | 72 | 69
units on a scale | -0.55 (1.039) | 1.45 (1.025) | -1.29 (1.056)
Statistical Analysis 1: Comparison: Placebo vs RVT-101 35 mg; Test type: Superiority; p = 0.158, Mixed Models Analysis — The threshold for statistical significance was p=0.05; Mean Difference (Final Values) = -2.01, 95% CI 2-sided [-4.80 to 0.79] — Placebo - active
Statistical Analysis 2: Comparison: Placebo vs RVT-101 70 mg; Test type: Superiority; p = 0.6069, Mixed Models Analysis — The threshold for statistical significance was p=0.05; Mean Difference (Final Values) = 0.74, 95% CI 2-sided [-2.08 to 3.55] — Placebo - active

2. Secondary Outcome: Alzheimer's Disease Assessment Scale - Cognitive Subscale 11 Items (ADAS-Cog-11) Change From Baseline at Week 24
Description: The 11-item ADAS-Cog assesses a range of cognitive abilities including memory, comprehension, orientation in time and place, and spontaneous speech. The ADAS-Cog-11 total score range is from 0 to 70, with a higher score indicating more severe cognitive impairment.
Time Frame: Change from Baseline at 24 weeks
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | RVT-101 35 mg | RVT-101 70 mg
Number analyzed (Participants) | 73 | 73 | 71
units on a scale | 1.68 (0.774) | 2.15 (0.769) | 1.01 (0.796)
Statistical Analysis 1: Comparison: Placebo vs RVT-101 35 mg; Test type: Superiority; p = 0.6531, Mixed Models Analysis; Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-2.55 to 1.60] — Placebo - active
Statistical Analysis 2: Comparison: Placebo vs RVT-101 70 mg; Test type: Superiority; p = 0.5274, Mixed Models Analysis — The threshold for statistical significance was p=0.05; Mean Difference (Final Values) = 0.67, 95% CI 2-sided [-1.41 to 2.75] — Placebo - active

3. Secondary Outcome: Clinician's Interview-Based Impression of Change Plus Caregiver Input (CIBIC+) Change From Baseline at Week 24
Description: To assess the effects of RVT-101 versus placebo on global function as measured by the Clinician's Interview-Based Impression of Change Plus Caregiver Input (CIBIC+) after 24 weeks of treatment. CIBIC+ is recorded on a 7-point scale with a score of 4 indicating no change, scores above 4 indicating worsening, and scores below 4 indicating improvement.
Time Frame: Change from Baseline at 24 weeks
Population: ITT Population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | RVT-101 35 mg | RVT-101 70 mg
Number analyzed (Participants) | 75 | 74 | 72
units on a scale | 4.42 (0.127) | 4.27 (0.128) | 4.35 (0.131)
Statistical Analysis 1: Comparison: Placebo vs RVT-101 35 mg; Test type: Superiority; p = 0.3953, Mixed Models Analysis — The threshold for statistical significance was p=0.05; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.2 to 0.5] — Placebo - active
Statistical Analysis 2: Comparison: Placebo vs RVT-101 70 mg; Test type: Superiority; p = 0.7008, Mixed Models Analysis — The threshold for statistical significance was p=0.05; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.28 to 0.42] — Placebo - active

ADVERSE EVENTS:
Time Frame: Screening through post treatment (up to 33 weeks)
Arm/Group | Placebo | RVT-101 35 mg | RVT-101 70 mg
All-Cause Mortality (participants affected / at risk) | 1/91 | 1/89 | 2/88
Serious Adverse Events (participants affected / at risk) | 11/91 | 11/89 | 13/88
Other Adverse Events (participants affected / at risk) | 66/91 | 69/89 | 59/88
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=91) | RVT-101 35 mg (N=89) | RVT-101 70 mg (N=88)
Deep vein Thrombosis (Vascular disorders) | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Atrial Flutter (Cardiac disorders) | 0 | 1 | 0
Trifascicular block (Cardiac disorders) | 0 | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Prostatic adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1 | 1
Dementia (Nervous system disorders) | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Delirium (Psychiatric disorders) | 2 | 0 | 0
Depression (Psychiatric disorders) | 0 | 1 | 0
Hallucination, visual (Psychiatric disorders) | 0 | 0 | 1
Mental status change (Psychiatric disorders) | 1 | 0 | 0
Neuropsychiatric syndrome (Psychiatric disorders) | 0 | 0 | 1
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 1
Enteritis (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 1
Volvulus (Gastrointestinal disorders) | 0 | 1 | 0
Cholecystitiis acute (Hepatobiliary disorders) | 1 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2
Sepsis (Infections and infestations) | 1 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=91) | RVT-101 35 mg (N=89) | RVT-101 70 mg (N=88)
Fall (Injury, poisoning and procedural complications) | 19 | 17 | 18
Urinary tract infection (Infections and infestations) | 4 | 7 | 7
Constipation (Gastrointestinal disorders) | 5 | 9 | 6
Orthostatic hypotension (Vascular disorders) | 12 | 3 | 5
Nasopharygitis (Respiratory, thoracic and mediastinal disorders) | 7 | 8 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 7 | 5
Hallucination, visual (Psychiatric disorders) | 4 | 6 | 3
Confusional state (Psychiatric disorders) | 3 | 5 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 7 | 5
Dizziness (Nervous system disorders) | 4 | 3 | 5
Nausea (Gastrointestinal disorders) | 2 | 4 | 5
Upper respiratory tract infection (Infections and infestations) | 6 | 3 | 2
Anxiety (Psychiatric disorders) | 3 | 5 | 2
Hypertension (Vascular disorders) | 5 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All proposed manuscripts, publications or abstracts must be reviewed and approved by the Sponsor 60 days prior to submission for publication. All confidential information identified by the Sponsor must be deleted prior to submission.

DOCUMENTS (2):
  • Study Protocol (2017-11-15): https://cdn.clinicaltrials.gov/large-docs/33/NCT02669433/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-14): https://cdn.clinicaltrials.gov/large-docs/33/NCT02669433/SAP_001.pdf